CLINICAL TRIAL: NCT01172509
Title: Transcranial Magnetic Stimulation (TMS) Measures of Plasticity and Excitatory/Inhibitory Ratio as Biomarkers for R-baclofen Effects in Normal Volunteers
Brief Title: TMS Measures of Plasticity and Excitatory/Inhibitory Ratio as Biomarkers: R-baclofen Effects in Normal Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: too much variability in the TMS measures
Sponsor: Gonzalez-Heydrich, Joseph, M.D. (Individual)
Collaborators: Boston Children's Hospital (Other); Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TMS_biomarker_Rbac_normals1
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Autism
Keywords: plasticity; excitatory; inhibitory; synaptic plasticity; R-Baclofen; TMS; transcranial magnetic stimulation; biomarker; autism
MeSH Terms: conditions — Autistic Disorder | interventions — arbaclofen placarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- sugar pill (Placebo Comparator): placebo administered under double blind conditions
  Interventions: Drug: R-baclofen
- 3 mg of R-baclofen (Experimental): 3 mg of R-Baclofen administered double blind
  Interventions: Drug: R-baclofen
- 10 mg of R-baclofen (Experimental): 10 mg of R-baclofen administered double-blind
  Interventions: Drug: R-baclofen
- 25 mg of R-baclofen (Experimental): 25 mg of R-baclofen administered double blind
  Interventions: Drug: R-baclofen
- second sugar pill (Placebo Comparator): the second placebo administered double blind
  Interventions: Drug: R-baclofen

INTERVENTIONS:
Drug: R-baclofen — oral R-baclofen at 0x2, 3, 10, and 25 mg
  Other Names: arbaclofen

SUMMARY:
Our overall objective is to apply Transcranial Magnetic Stimulation (TMS) to develop measures of human synaptic plasticity and of brain excitatory:inhibitory ratio (E:I ratio), which we propose as novel biomarkers and outcome measures that will expedite clinical trials of treatments for Autism Spectrum Disorder (ASD). One potential therapeutic agent, R-baclofen will be investigated under this protocol.

TMS is a safe, inexpensive and noninvasive means to focally stimulate the human brain. Presently, TMS is in extensive use as a means to measure regional brain excitability, which is dependent on local synaptic strength. TMS can be used to temporarily alter synaptic strength as well as to acutely measure levels of cortical excitability and short and long interval inhibition. Since altered synaptic plasticity and an imbalanced inhibitory:excitatory ratio are cited as fundamental abnormalities in ASD, we hypothesize that both severity of ASD-related learning deficits and their improvement after therapy will correlate with TMS measures of synaptic plasticity and E:I ratio. We propose to embed TMS measures of synaptic plasticity and E:I ratio in a 'Proof of Principal' trial of R-baclofen and to examine:

Aim 1: Whether R-baclofen (a potential therapeutic agent for ASD) predictably alters TMS measures of synaptic plasticity and E:I ratio as a function of plasma concentration in adult volunteers. We will test the following hypotheses:

1. R-baclofen produces a significant change in TMS measures of LTD and E:I ratio; and
2. R-baclofen plasma levels and TMS measures of LTD and E:I ratio show a predictable exposure-response relationship.

Exploratory Aim 1: Whether the presence of genetic polymorphisms of the BDNF and GABA-B receptor genes has a moderating effect on TMS measures and on R-baclofen effects. We will test the following hypotheses:

1. Presence of the BDNF val66met allele will be associated with decreased long-term depression (LTD) of cortical excitability
2. Polymorphisms of GABA-B receptor genes will be associated with altered magnitude of response to R-baclofen as measured by TMS

DETAILED DESCRIPTION:
The design is a double-blind placebo controlled 5 way crossover trial of a single dose each of placebo x 2 (0 mg), 3, 10, and 25 mg of R-baclofen followed by plasma levels at 0, 30, 60, 90, and 140 minutes after each dose; and TMS testing at 0, 30, 60, 90 (cTBS application at 90 minute time point), 95, and then periodically every 5-10 minutes until the MEPs return to baseline. There will be a total of 7 visits. Patients will come in for a screening visit, then scheduled to return for 1 baseline visit (cTBS without drug) and 5 crossover visits. At each crossover visit a venous line will be placed for blood sampling and a single dose of study drug at one of the five dose levels will be given orally at time 0. There will be a one-week washout between each of the crossover arms (R-baclofen has a mean Tmax of approximately 80 minutes and a terminal half life of 4.9 hour).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30
* IQ: higher than 85
* Normal physical examination

Exclusion Criteria

* significant medical problems
* ongoing medications
* All female participants are required to have a negative pregnancy test

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
percent of baseline TMS-induced measures of (1) human synaptic plasticity (LTD) | at 90 minutes after study drug dose
  Synaptic plasticity or LTD will be measured using the MEP in response to stimulation set at 80% of the active motor threshold. This MEP will be measured at 90 minutes after study drug dose to establish baseline MEP amplitude then LTD will be induced with the cTBS procedure. The amount of LTD remaining at the different time points, post-cTBS will be quantified by measuring the MEPs and dividing it by the baseline MEP. This will yield a percent of baseline MEP at the various time points.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gonzalez-Heydrich, MD, Study Director — Boston Children's Hospital; Alvaro Pascual-Leone, M.D. Ph. D., Study Chair — Berenson-Allen Center for Noninvansive Brain Stimulation BIDMC; Lindsay M Oberman, Ph. D, Principal Investigator — Berenson-Allen Center for Noninvansive Brain Stimulation BIDMC
Locations (1):
- Berenson-Allen Center for Noninvansive Brain Stimulation Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States